CLINICAL TRIAL: NCT00994422
Title: A Double-Blind Randomized Study to Compare the Safety, Local Tolerability and Efficacy of a 0.5% Ivermectin Cream Compared to a Topical Vehicle Control in Subjects With Pediculus Humanus Capitis Infestation
Brief Title: Study Comparing the Safety and Efficacy of 0.5% Ivermectin Cream to Placebo in Lice Infested Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Topaz Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOP010
Record Dates: First submitted 2009-10-09; First posted 2009-10-14 (Estimated); Results first posted 2012-04-04 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Head Lice
Keywords: PEDICULUS HUMANUS CAPITIS; Head Lice

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.5% ivermectin cream (Experimental)
  Interventions: Drug: Ivermectin cream
- vehicle control (Placebo Comparator)
  Interventions: Drug: vehicle control

INTERVENTIONS:
Drug: Ivermectin cream — Up to 4 ounces of topical 0.5% Ivermectin Cream applied to the hair and scalp on day 1.
  Arms: 0.5% ivermectin cream
Drug: vehicle control — Up to 4 ounces of vehicle control applied to the hair and scalp on day 1
  Arms: vehicle control

SUMMARY:
The purpose of this study is to compare the safety and efficacy of a 0.5% ivermectin cream to a placebo in subjects infested with head lice when used in an "at home" environment.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have an active head lice infestation defined as: At least 1 live louse (adult and/or nymph) present on the scalp and/or hair, as determined by a trained evaluator (with the exception of the male head of household who may self-assess as being lice free).
* Subject is male or female.
* Subject weighs at least 15kg (33 lbs).
* Subject is in good general health based on medical history.
* Each subject must have an appropriately signed Informed Consent agreement. A caregiver must sign an Informed Consent agreement for children not old enough to do so. Children of a specified age will be administered a child's assent form.
* The caregiver of a subject must be willing to allow all household members to be screened for head lice. If other household members are found to have an active head lice infestation, according to the criteria a (above), they must be willing and able to participate in the study. No more than one working male per family may be excluded from evaluation if he is self-assessed as being lice free and cannot come in due to his work schedule. If this individual may have lice, he must come to the test facility; otherwise the entire household will be excluded from study participation.
* Subject and/or their caregiver must be physically able and willing to apply the test article.
* Subject agrees not to use any other form of lice treatments (commercial, community-anecdotal, or mechanical/manual) while they are participating in the study.
* Following application and rinsing of Study Treatment, subject agrees not to shampoo, wash, or rinse their hair or scalp until the 24-hour post-treatment evaluation has been completed.
* Subject agrees that they will not cut or chemically treat their hair while they are participating in the study.
* Subject agrees to follow all study instructions.
* Female subjects of childbearing potential (including a female caregiver even if she is not being treated) must be willing to have a urine pregnancy test.
* In the event of a subject judged to be incapable of self-treating, the household must have a caregiver willing to apply the treatment at home.

Exclusion Criteria:

* History of irritation or sensitivity to ivermectin or the cream components, pediculicides or hair care products.
* Presentation at the treatment site with visible skin/scalp condition(s) that are not attributable to head lice infestation, such as an erythema score that is >2, blisters, vesicles which, in the opinion of the investigative personnel or sponsor, will interfere with safety and/or efficacy evaluations.
* Presentation at the treatment site with eczema or atopic dermatitis on the skin/scalp.
* Treatment with a marketed pediculicide (Over the counter [OTC] or Prescription) in the last 7 days.
* Any condition or illness that, in the opinion of the investigator, may compromise the objective of the protocol.
* Is receiving any other treatment which, in the opinion of the investigator or study monitor, may interfere with the study results.
* Females (including caregivers who come in contact with the investigational product) who are pregnant, nursing or planning a pregnancy. (NOTE: female caregivers and all enrolled females of childbearing potential must have a negative urine pregnancy test prior to treatment). If a household has a pregnant female who has an active case of lice, the entire household is excluded from participation. If this pregnant household member does not have an active infestation, this individual must NOT be the caregiver (one who provides treatment to other household members).
* Is of child-bearing potential and unwilling to use an adequate method of contraception for the duration of the study. Adequate methods of contraception include: abstinence, vasectomized partner, oral birth control pills, birth control injections or patches, Intra Uterine Devices, condoms with a spermicidal jelly or a diaphragm with spermicidal jelly, surgical sterilization.
* Participation in a previous investigational drug study within the past 30 days.
* Does not understand the requirements for study participation and/or may likely exhibit poor compliance, in the opinion of the investigator.
* Does not have a known household affiliation with their household members (i.e., do not stay in one household consistently, sleeping at one place several nights and then at another place or location). Household is defined as living in a shared area or space (for example the same house or apartment unit).

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Topaz
Locations (12):
- United States (12):
  - Cactus Kids Pediatrics, Yuma, Arizona
  - Impact Clinical Trials, Los Angeles, California
  - Lice Cleanique, LLC, Delray Beach, Florida
  - Hill-Top Research Corp, St. Petersburg, Florida
  - LSRN, West Palm Beach, Florida
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - Haywood Pediatric Adolescent Medicine Group, PA, Clyde, North Carolina
  - Hill Top Research Corp., Miamiville, Ohio
  - LSRN, Nashville, Tennessee
  - Northeast Houston Pediatric Clinic, Houston, Texas
  - Virgina Clinical Research, Inc., Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and treated from 13 October 2009 to 02 December 2009 in 12 US clinical centers.
Pre-assignment Details: A total of 247 of the 264 randomized participants who met the inclusion and exclusion criteria received treatment in the study.
Groups:
- 0.5% Ivermectin: Participants received a single application of Ivermectin cream on Day 1.
- Placebo (Vehicle Control): Participants received a single application of vehicle control cream on Day 1.
Period: Overall Study
Arm/Group | 0.5% Ivermectin | Placebo (Vehicle Control)
Started | 192 | 55
Completed | 185 | 54
Not Completed | 7 | 1
Not completed — Lost to Follow-up | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5% Ivermectin | Placebo (Vehicle Control) | Total
Number analyzed (Participants) | 192 | 55 | 247
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 147 | 35 | 182
  Between 18 and 65 years | 45 | 20 | 65
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 15.9 (12.9) | 19.6 (14.4) | 16.76 (13.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 42 | 203
  Male | 31 | 13 | 44
Region of Enrollment [Number; unit: Participants]
  United States | 192 | 55 | 247

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Success Following Treatment With Either Ivermectin or Placebo (Vehicle Control)
Description: Treatment success was defined as the absence of live lice and was determined by visual examination of hair and scalp by a trained evaluator.
Time Frame: Days 2 up to Day 15 post-treatment
Population: Treatment success was assessed in the Intent-to-treat population. Any participant with live lice on or after Day 2 received an FDA approved head lice treatment and was classified as a treatment failure, imputed as such for remaining assessments.
Measure: Number; unit: Percent of Participants
Arm/Group | 0.5% Ivermectin | Placebo (Vehicle Control)
Number analyzed (Participants) | 192 | 55
Percent of Participants
  Day 2 (N = 192, 55) | 95 | 53 [0 to 0]
  Day 8 (N = 191, 55) | 83 | 49 [0 to 0]
  Day 15 (N = 185, 54) | 76 | 35 [0 to 0]

2. Primary Outcome: Number of Participants Reporting Adverse Events Post-Treatment With Either Ivermectin or Placebo (Vehicle Control)
Time Frame: Day 1 up to Day 28 post-application
Population: Adverse events were assessed in the Intent-to-treat (Safety) population.
Measure: Number; unit: Participants
Groups:
- 0.5% Ivermectin: Participants received a single application of 0.5% ivermectin cream on Day 1.
- Vehicle Control: Participants received a single application of vehicle control cream on Day 1.
Arm/Group | 0.5% Ivermectin | Vehicle Control
Number analyzed (Participants) | 192 | 55
Participants
  Conjunctivitis | 1 | 0 [0 to 0]
  Application site pruritus | 1 | 1 [0 to 0]
  Influenza | 2 | 0 [0 to 0]
  Nail bed infection | 1 | 0 [0 to 0]
  Pharyngitis | 1 | 0 [0 to 0]
  Pyoderma | 1 | 0 [0 to 0]
  Swine influenza | 1 | 0 [0 to 0]
  Upper respiratory tract infection | 5 | 0 [0 to 0]
  Contusion | 1 | 0 [0 to 0]
  Excoriation | 8 | 4 [0 to 0]
  Scratch | 1 | 0 [0 to 0]
  Headache | 1 | 0 [0 to 0]
  Asthma | 1 | 0
  Dyspnoea | 1 | 0
  Oropharyngeal pain | 2 | 0
  Erythema | 2 | 1
  Pruritus | 4 | 0
  Rash maculo-papular | 1 | 0

3. Primary Outcome: Summary of the Reported Skin/Scalp Irritations Before and Post-treatment With Either Ivermectin or Placebo (Vehicle Control)
Description: Participants skin/scalp irritations were assessed before treatment (Day 1) and Post-treatment with either Ivermectin or placebo by a trained evaluator.
  Severe scalp irritations were defined as follows:
  Severe Pruritus - Nearly constant, frequent scratching, very bothersome; Severe Erythema - Large areas of the scalp are red; Severe Excoriation: Widespread breaking of the skin involving most of the scalp; Severe Pyoderma - Lesions with crusting or other evidence of infection, involving most of the scalp.
Time Frame: Day 1 up to Day 15 post-application
Population: Local tolerability was assessed in the Intent-to-treat (Safety) population.
Measure: Number; unit: Participants
Arm/Group | 0.5% Ivermectin | Vehicle Control
Number analyzed (Participants) | 192 | 55
Participants
  Any Erythema Day 1 (Pre-treatment; N = 192, 55) | 26 | 5 [0 to 0]
  Severe Erythema Day 1 (Pre-treatment; N = 192, 55) | 0 | 0 [0 to 0]
  Any Erythema Day 2 (N = 192, 55) | 18 | 3 [0 to 0]
  Severe Erythema Day 2 (N = 192, 55) | 0 | 0 [0 to 0]
  Any Erythema Day 8 (N = 181, 29) | 7 | 0 [0 to 0]
  Severe Erythema Day 8 (N = 181, 29) | 0 | 0 [0 to 0]
  Any Erythema Day 15 (N = 152, 26) | 3 | 0 [0 to 0]
  Severe Erythema Day 15 (N = 152, 26) | 0 | 0 [0 to 0]
  Any Excoriation Day 1 (Pre-treatment; N = 192, 55) | 31 | 7 [0 to 0]
  Severe Excoriation Day 1 (Pre-treatment; N=192, 55 | 0 | 0 [0 to 0]
  Any Excoriation Day 2 (N = 192, 55) | 27 | 7 [0 to 0]
  Severe Excoriation Day 2 (N = 192, 55) | 0 | 0 [0 to 0]
  Any Excoriation Day 8 (N = 181, 29) | 15 | 2 [0 to 0]
  Severe Excoriation Day 8 (N = 181, 29) | 0 | 0 [0 to 0]
  Any Excoriation Day 15 (N = 152, 26) | 4 | 0 [0 to 0]
  Severe Excoriation Day 15 (N = 152, 26) | 0 | 0 [0 to 0]
  Any Pruritus Day 1 (Pre-treatment; N = 192, 55) | 134 | 36 [0 to 0]
  Severe Pruritus Day 1 (Pre-treatment; N = 192, 55) | 17 | 3 [0 to 0]
  Any Pruritus Day 2 (N = 192, 55) | 56 | 25 [0 to 0]
  Severe Pruritus Day 2 (N = 192, 55) | 0 | 0 [0 to 0]
  Any Pruritus Day 8 (N = 181, 29) | 32 | 5 [0 to 0]
  Severe Pruritus Day 8 (N = 181, 29) | 0 | 0 [0 to 0]
  Any Pruritus Day 15 (N = 152, 26) | 8 | 2 [0 to 0]
  Severe Pruritus Day 15 (N = 152, 26) | 0 | 0 [0 to 0]
  Any Pyoderma Day 1 (Pre-treatment, N = 192, 55) | 1 | 1 [0 to 0]
  Severe Pyoderma Day 1 (Pre-treatment; N = 192, 55) | 0 | 0 [0 to 0]
  Any Pyoderma Day 2 (N = 192, 55) | 1 | 1 [0 to 0]
  Severe Pyoderma Day 2 (N = 192, 55) | 0 | 0 [0 to 0]
  Any Pyoderma Day 8 (N = 181, 29) | 1 | 0 [0 to 0]
  Severe Pyoderma Day 8 (N = 181, 29) | 0 | 0 [0 to 0]
  Any Pyoderma Day 15 (N = 152, 26) | 0 | 0 [0 to 0]
  Severe Pyoderma Day 15 (N = 152, 26) | 0 | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected form Day 1 up to Day 28 post-treatment with either Ivermectin or Placebo
Arm/Group | 0.5% Ivermectin | Placebo (Vehicle Control)
Serious Adverse Events (participants affected / at risk) | 0/192 | 0/55
Other Adverse Events (participants affected / at risk) | 8/192 | 4/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.5% Ivermectin (N=192) | Placebo (Vehicle Control) (N=55)
Excoriation (Injury, poisoning and procedural complications) | 8 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications